CLINICAL TRIAL: NCT04851574
Title: Optimization of Rocuronium and Sugammadex Dosing Based on Their Pharmacokinetic and Pharmacodynamic (PKPD) Profile in Children Undergoing General Anesthesia
Brief Title: PKPD of Rocuronium and Sugammadex Profile in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Agnieszka Bienert, Full Professor, Poznan University of Medical Sciences
Other Study IDs: 161/2017
Record Dates: First submitted 2021-03-07; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: General Anesthetic Drug Adverse Reaction
Keywords: General anesthesia; Children
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group I with dose of Sugammadex of 0.5 Mg/kg: After general anesthesia children received one dose of 0.5 Mg/kg of Sugammadex to reverse neuromuscular blockade.
  Interventions: Drug: Sugammadex Injection
- Group II with dose of Sugammadex of 1.0 Mg/kg: After general anesthesia children received one dose of 1.0 Mg/kg of Sugammadex to reverse neuromuscular blockade.
  Interventions: Drug: Sugammadex Injection
- Group III with dose of Sugammadex of 2.0 Mg/kg: After general anesthesia children received one dose of 2.0 Mg/kg of Sugammadex to reverse neuromuscular blockade.
  Interventions: Drug: Sugammadex Injection

INTERVENTIONS:
Drug: Sugammadex Injection — Sugammadex was administered in the dose of 0.5 Mg/kg or 1.0 Mg/kg or 2.0 Mg/kg to reverse neuromuscular blockade.
  Other Names: Sugammadex 100Mg/ml Intravenous Solution

SUMMARY:
The aim of the study is to assess the pharmacokinetic and pharmacodynamic properties of rocuronium and sugammadex and their clinical effect in the terms of both the relaxation of paralysed muscles (rocuronium) and the reversal of neuromuscular blockade (sugammadex) in children over 2 years of age undergoing general anesthesia for surgical procedures needing muscle relaxation for more than 30 minutes.

DETAILED DESCRIPTION:
The study group was divided into three subgroups depending on the different doses of sugammadex. Group I received dose of 0.5 Mg/kg, Group II - 1.0 Mg/kg and Group III received dose of 2 Mg/kg of sugammadex. General anesthesia was performed among all included patients at the same way. During general anesthesia monitoring of TOF - Train-of-four, was used to assess the muscle relaxation force of rocuronium as well as the reversal of neuromuscular blockade by sugammadex. For this purpose, 1.5 ml of blood samples taken 8 times, were collected to determine the PKPD of the tested drugs, according to own protocol.

ELIGIBILITY:
Inclusion Criteria:

* age 2-18 years
* ASA I-II
* qualification to surgival procedures requiring muscle relaxation for more than 30 minutes
* parental consent of children below 16 yrs and parental and child's consent if child was older than 16 yrs of age
* Bioethical Commission approvement No 161/17

Exclusion Criteria:

* ASA III and more
* age below 2 yrs
* lack of consent
* allergy to studied drugs
* less than 30 minutes of relaxation required

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, aged 2-18 yrs, assessed according to American Society of Anesthesiologists (ASA) scale as I or II, qualified to surgical procedures requiring muscle relaxation for more than 30 minutes, and undergoing general anesthesia
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Recovery of muscular contraction following sugammadex injection | up to 24 hours
  Recovery of muscular contraction following sugammadex in reversal of neuromuscular blockade in children

SECONDARY OUTCOMES:
Sugammadex serum concentration [ng/ml] | up to 24 hours
  Different doses of Sugammadex have influence on the pharmacokinetic and pharmacodynamic profile
Heart rate [beats per minute] | up to 24 hours
  Measurement of the heart rate during and after anesthesia
Systolic blood pressure [mmHg] | up to 24 hours
  Measurement of the systolic blood pressure during and after anesthesia
Diastolic blood pressure [mmHg] | up to 24 hours
  Measurement of the diastolic blood pressure during and after anesthesia
Blood Oxygen Saturation [percent] | up to 24 hours
  Measurement of the blood oxygen saturation during and after anesthesia
Train-of-four monitoring | through study completion
  Standard practice evaluation of muscle strength during anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Bartkowska-Sniatkowska, MD PhD, Study Chair — Department of Pediatric Anesthesiology and Intensive Care
Locations (1):
- Alicja Bartkowska-Sniatkowska, Poznan, Grand Poland, Poland

IPD SHARING:
Plan to Share IPD: Yes
PK and PD data (concentration/effect/time profiles) of individuals will be available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available in 4-6 months and available for 5 years
Access Criteria: Scientists

REFERENCES:
- [Derived] Grzeskowiak M, Bienert A, Wiczling P, Malec M, Grzelak J, Jarosz K, Ber J, Ksiazkiewicz M, Rosada-Kurasinska J, Grzeskowiak E, Bartkowska-Sniatkowska A. Population Pharmacokinetic-Pharmacodynamic Modeling and Probability of Target Attainment Analysis of Rocuronium and Sugammadex in Children Undergoing Surgery. Eur J Drug Metab Pharmacokinet. 2023 Jan;48(1):101-114. doi: 10.1007/s13318-022-00809-1. Epub 2022 Dec 8. PMID 36477706